CLINICAL TRIAL: NCT02030379
Title: Developing an Online Clinical Trial Specific Question Prompt List
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-14970; HM14970 (Other: VCU Institutional Review Board)
Record Dates: First submitted 2013-12-10; First posted 2014-01-08 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Online QPL-CT to Oncologist (Experimental): Use the online QPL-CT to prioritize their questions and the prioritized list will be conveyed to their oncologist
  Interventions: Behavioral: QPL-CT
- Online QPL-CT (Experimental): Use the online QPL-CT to prioritize their questions.
  Interventions: Behavioral: QPL-CT
- Pencil and Paper QPL-CT (Experimental): Use pencil and paper QPL-CT to prioritize their questions
  Interventions: Behavioral: QPL-CT

INTERVENTIONS:
Behavioral: QPL-CT — Use the QPL-CT to prioritize questions

SUMMARY:
The investigators will leverage e-technologies to provide an online version of the Question Prompt LIst (QPL-CT), that patients access via available iPads, enabling both the real-time prioritizing of patient questions as well as the seamless delivery of these questions to their treating physician (and other members of their clinical team) via the VCU Health System (VCUHS) patient portal, and the electronic medical record (EMR) prior to a consultation to discuss a clinical trial

DETAILED DESCRIPTION:
The investigators propose to conduct pilot work to inform our knowledge of optimal methods of utilizing QPLs and will use the QPL-CT as an example. The investigators will leverage e-technologies to provide an online version of the QPL-CT, that patients access via available iPads, enabling both the real-time prioritizing of patient questions as well as the seamless delivery of these questions to their treating physician (and other members of their clinical team) via the VCU Health System (VCUHS) patient portal, and the EMR prior to a consultation to discuss a clinical trial. The investigators will use a pilot randomized clinical trial design to demonstrate the efficacy of the online QPL-CT versus a paper and pencil QPL-CT to increase question asking, patient understanding of trial information and reduce patients conflict over their upcoming decision to join a trial

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Fluent in English
* eligible for a therapeutic clinical trial
* Patients of recruited oncologists

Exclusion Criteria:

* Healthy subjects
* Not eligible for a therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Online QPL-CT to Oncologist | 30 days
  Use online QPL-CT to prioritize their questions and the prioritized list will be conveyed to their oncologist. Investigators will evaluate the efficacy of the online QPL-CT to increase question asking, patient understanding of trial information and reduce patients conflict over their upcoming decision to join a trial.

SECONDARY OUTCOMES:
Impact of providing physicians patient's QPL-CT | 30 days
  Examine the impact of providing physicians their patient's prioritized QPL-CT on information provision and decision making process as measured by the Decision Analysis System for Oncology

OTHER OUTCOMES:
Test the feasibility of using the online QPL-CT for patients and physicians | 30 days
  Patients will complete an exit interview at the completion of patient's consultation asking about the patient's impressions of the online QPL-CT including its ease of use and the patient's perceptions of its influence on consultation communication. Physicians will complete a brief interview on one occasion at the completion of patient recruitment asking about the impact of the prioritized QPL-CT on consultation communication.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States